CLINICAL TRIAL: NCT03901326
Title: The Effect of On-site CT-derived Fractional Flow Reserve on the Management Making for the Patients With Stable Chest Pain (TARGET Trial)
Brief Title: Role of On-site CT-derived FFR in the Management of Suspect CAD Patients
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Qilu Hospital of Shandong University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yundai Chen, Director of Cardiology Department, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2019-025-01
Record Dates: First submitted 2019-03-30; First posted 2019-04-03 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coronary computed tomographic angiography; Fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTA/CT-FFR care group (Experimental): If the subjects are randomly allocated to CT-FFR arm, they will be examined by on-site DeepFFR for three major epicardial coronary arteries. If the result of CT-FFR calculation is less than or equal to 0.8 in one or more major coronary arteries, the patient will be referred to ICA directly; if the result of CT-FFR value is more than 0.8, optimal medical therapy will be recommended. The decision on the mode of revascularization is left to the treating cardiologists and depends on local practice standard.
  Interventions: Diagnostic Test: CT-FFR assessment
- Routine clinically-indicated diagnostic care group (No Intervention): If the subjects are randomized to usual care arm, attending physicians will decide the next step of diagnosis and treatment, such as exercise ECG, stress cardiac echo, cardiac MR, and SPECT. According to the results of examination combined with risk factors assessment and clinical manifestations, physicians should provide recommendation whether the subjects would undergo ICA or not.

INTERVENTIONS:
Diagnostic Test: CT-FFR assessment — When subjects are randomized to the CTA/CT-FFR arm, FFR based on the coronary CTA imaging will be measured. DEEPVESSEL FFR workstation is very dedicated software utilizing the original CTA imaging to meter simulated FFR values based on a machine learning algorithm. The first step is to extract a 3D coronary artery model and generate coronary centerlines which are similar to the routine reconstruction of coronary CTA. The centerlines are extracted using a minimal path extraction filter. Then a novel path-based deep learning model, referred to DEEPVESSEL FFR, is used to predict the simulated FFR values on the vascular centerlines. Deep learning algorithm is used to establish characteristic sample database of coronary hemodynamics characteristic parameters. When deep training model is proved to be valid, it is applied to a new lesion-specific measurement. Lesion-specific CT-FFR is defined as simulated FFR value at distance of 20mm away from the lesion of interest.
  Arms: CTA/CT-FFR care group

SUMMARY:
The primary of this registry is to evaluate whether the availability of CTA/CT-FFR procedure could effectively optimize the flow of clinical practice of stable chest pain versus conventional clinical pathway in decision making, avoid the overuse of invasive procedure, finally improve clinical prognosis and reduce total medical expenditure. This registry is randomized, open labeled, prospective designed and will be performed in 6 Chinese hospitals. Approximately 1200 subjects will be enrolled and subsequently assigned to either routine clinically-indicated diagnostic care group (CID arm) or CTA/CT-FFR care group (CTA/CT-FFR arm) via computer-generated random numbers (1:1 ratio)

DETAILED DESCRIPTION:
Based on the clinical fact that less stress myocardial perfusion scan are performed rather than stress exercise electrocardiogram (ECG) in China, more patients undergo coronary computed tomographic angiography (CTA) for determining whether they should be sent to catheter lab. However, nearly 30% of patients sent to catheter lab were found without obstructive coronary artery disease (CAD) and this invasive procedure was unnecessary and overused partly. Fortunately, fractional flow reserve (FFR) based non-invasive CT algorithm technology (CT-FFR) showed a great potential in detecting functional myocardial ischemia related to coronary specific lesion (Discovery-Flow, DEFACTO and NXT trial)[1-3]. Moreover, clinical care guided by CT-FFR could provide benefits with equivalent clinical outcomes and lower expenditure, compared with routine clinical care over 1-year follow-up (Platform trial). On the other aspect, ADVANCE trial revealed that CT-FFR modified treatment recommendation was associated with less negative invasive coronary angiography (ICA), predicted revascularization and identified subjects at low risk of adverse events through 90 days in real-world. However, these studies was not randomized designed and selection bias still existed. So our trial aims to evaluate whether CTA/CT-FFR outperforms the regular diagnostic care in ruling out patients without significantly obstructive CAD before catheter lab and improving clinical prognosis during follow-up in a randomized design.

ELIGIBILITY:
Inclusion Criteria:

* New-onset chest pain suspicious for CAD
* Coronary CTA result showed that the diameter stenosis is between 30 and 90% in at least one major coronary artery (coronary artery diameter ≥ 2.5 mm)
* Intermediate-to-high pretest probability of CAD based on CAD Consortium Score
* No prior evaluation for this episode of symptoms
* Agree to participate in this clinical study and sign written informed consent

Exclusion Criteria:

* Diagnosed or suspected acute coronary syndrome requiring hospitalization or emergent testing
* Hemodynamically or clinically unstable condition systolic blood pressure < 90 mmHg or serious atrial or ventricular arrhythmias
* Known CAD with prior myocardial infarction, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG), or any angiographic evidence of ≥ 50% stenosis in any major coronary artery
* Patients with left main branch stenosis ≥ 50% or major coronary artery stenosis > 90%
* Known severe congenital, valvular (moderate and above), or cardiomyopathy process (hypertrophic cardiomyopathy or reduced systolic left ventricular function ≤ 40%) which could explain cardiac symptoms
* Unable to provide written informed consent or participate in long-term follow-up.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1216 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Ph.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711
- [Background] Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S; NXT Trial Study Group. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014 Apr 1;63(12):1145-1155. doi: 10.1016/j.jacc.2013.11.043. Epub 2014 Jan 30. PMID 24486266
- [Background] Douglas PS, De Bruyne B, Pontone G, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C, Hlatky MA; PLATFORM Investigators. 1-Year Outcomes of FFRCT-Guided Care in Patients With Suspected Coronary Disease: The PLATFORM Study. J Am Coll Cardiol. 2016 Aug 2;68(5):435-445. doi: 10.1016/j.jacc.2016.05.057. PMID 27470449
- [Background] Fairbairn TA, Nieman K, Akasaka T, Norgaard BL, Berman DS, Raff G, Hurwitz-Koweek LM, Pontone G, Kawasaki T, Sand NP, Jensen JM, Amano T, Poon M, Ovrehus K, Sonck J, Rabbat M, Mullen S, De Bruyne B, Rogers C, Matsuo H, Bax JJ, Leipsic J, Patel MR. Real-world clinical utility and impact on clinical decision-making of coronary computed tomography angiography-derived fractional flow reserve: lessons from the ADVANCE Registry. Eur Heart J. 2018 Nov 1;39(41):3701-3711. doi: 10.1093/eurheartj/ehy530. PMID 30165613
- [Background] Norgaard BL, Hjort J, Gaur S, Hansson N, Botker HE, Leipsic J, Mathiassen ON, Grove EL, Pedersen K, Christiansen EH, Kaltoft A, Gormsen LC, Maeng M, Terkelsen CJ, Kristensen SD, Krusell LR, Jensen JM. Clinical Use of Coronary CTA-Derived FFR for Decision-Making in Stable CAD. JACC Cardiovasc Imaging. 2017 May;10(5):541-550. doi: 10.1016/j.jcmg.2015.11.025. Epub 2016 Apr 13. PMID 27085447
- [Background] Colleran R, Douglas PS, Hadamitzky M, Gutberlet M, Lehmkuhl L, Foldyna B, Woinke M, Hink U, Nadjiri J, Wilk A, Wang F, Pontone G, Hlatky MA, Rogers C, Byrne RA. An FFRCT diagnostic strategy versus usual care in patients with suspected coronary artery disease planned for invasive coronary angiography at German sites: one-year results of a subgroup analysis of the PLATFORM (Prospective Longitudinal Trial of FFRCT: Outcome and Resource Impacts) study. Open Heart. 2017 Mar 22;4(1):e000526. doi: 10.1136/openhrt-2016-000526. eCollection 2017. PMID 28674617
- [Background] Collet C, Onuma Y, Andreini D, Sonck J, Pompilio G, Mushtaq S, La Meir M, Miyazaki Y, de Mey J, Gaemperli O, Ouda A, Maureira JP, Mandry D, Camenzind E, Macron L, Doenst T, Teichgraber U, Sigusch H, Asano T, Katagiri Y, Morel MA, Lindeboom W, Pontone G, Luscher TF, Bartorelli AL, Serruys PW. Coronary computed tomography angiography for heart team decision-making in multivessel coronary artery disease. Eur Heart J. 2018 Nov 1;39(41):3689-3698. doi: 10.1093/eurheartj/ehy581. PMID 30312411
- [Background] Norgaard BL, Terkelsen CJ, Mathiassen ON, Grove EL, Botker HE, Parner E, Leipsic J, Steffensen FH, Riis AH, Pedersen K, Christiansen EH, Maeng M, Krusell LR, Kristensen SD, Eftekhari A, Jakobsen L, Jensen JM. Coronary CT Angiographic and Flow Reserve-Guided Management of Patients With Stable Ischemic Heart Disease. J Am Coll Cardiol. 2018 Oct 30;72(18):2123-2134. doi: 10.1016/j.jacc.2018.07.043. Epub 2018 Aug 25. PMID 30153968
- [Background] Jensen JM, Botker HE, Mathiassen ON, Grove EL, Ovrehus KA, Pedersen KB, Terkelsen CJ, Christiansen EH, Maeng M, Leipsic J, Kaltoft A, Jakobsen L, Sorensen JT, Thim T, Kristensen SD, Krusell LR, Norgaard BL. Computed tomography derived fractional flow reserve testing in stable patients with typical angina pectoris: influence on downstream rate of invasive coronary angiography. Eur Heart J Cardiovasc Imaging. 2018 Apr 1;19(4):405-414. doi: 10.1093/ehjci/jex068. PMID 28444153
- [Derived] Yang J, Shan D, Wang X, Sun X, Shao M, Wang K, Pan Y, Wang Z, Schoepf UJ, Savage RH, Zhang M, Dong M, Xu L, Zhou Y, Ma X, Hu X, Xia L, Zeng H, Liu Z, Chen Y. On-Site Computed Tomography-Derived Fractional Flow Reserve to Guide Management of Patients With Stable Coronary Artery Disease: The TARGET Randomized Trial. Circulation. 2023 May 2;147(18):1369-1381. doi: 10.1161/CIRCULATIONAHA.123.063996. Epub 2023 Mar 4. PMID 36870065
- [Derived] Yang J, Shan D, Dong M, Wang Z, Ma X, Hu X, Zeng H, Chen Y. The effect of on-site CT-derived fractional flow reserve on the management of decision making for patients with stable chest pain (TARGET trial): objective, rationale, and design. Trials. 2020 Aug 20;21(1):728. doi: 10.1186/s13063-020-04649-9. PMID 32819429

RESULTS

PARTICIPANT FLOW:
Groups:
- CTA/CT-FFR Care Group: If the subjects are randomly allocated to CT-FFR arm, they will be examined by DeepFFR for three major epicardial arteries. If the result of CT-FFR calculation is less than or equal to 0.8 in one or more major，coronary arteries, the patient will be referred to ICA directly; if the result of CT-FFR value is more than 0.8, optimal medical therapy will be recommended. The decision on the mode of revascularization is left to the treating cardiologists and depends on local practice standard.
  CT-FFR: DeepFFR workstation is very dedicated software utilizing the original CTA imaging to meter simulated FFR values in artificial intelligence model.The first step is to extract a 3D coronary artery model and generate coronary centerlines which are similar to the routine reconstruction of coronary CTA. The centerlines are extracted using a minimal path extraction filter. Then a novel path-based deep learning model, referred to DeepFFR, is used to predict the simulated FFR values on the vascular centerlines. Deep learning algorithm is used to establish characteristic sample database of coronary hemodynamics characteristic parameters. When deep training model is proved to be valid, it is applied to a new lesion-specific measurement. Lesion-specific CT-FFR is defined as simulated FFR value at distance of 20mm away from the lesion of interest.
Period: Overall Study
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group
Started | 608 | 608
Completed | 608 | 608
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group | Total
Number analyzed (Participants) | 608 | 608 | 1216
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (8.3) | 59.2 (11.5) | 59.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 221 | 431
  Male | 398 | 387 | 785
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Median (Inter-Quartile Range); unit: kg/m²] | 25.1 [23.3 to 27.8] | 25.3 [23.0 to 27.3] | 25.2 [23.3 to 27.6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ICA Without Obstructive CAD or Intervention
Description: Number of those patients with planned ICA in whom no significant obstructive CAD (no stenosis≥70% by core lab quantitative analysis or invasive FFR≤0.8) is found or interventions (including stent implantation, balloon dilation and bypass graft) are performed during ICA within 90 days.
Time Frame: 90 days
Population: In the general population, patients with severe coronary stenosis maybe considered to be sent to catheter room, while the main endpoint is the negative findings during angiography. Therefore, for instance, the total population in the CT-FFR group is 608 (row1), of which 421 patients (row2, 3) enter the catheter room for coronary angiography. Therefore, the proportion of the three rows is different.
Measure: Count of Participants; unit: Participants
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group
Number analyzed (Participants) | 608 | 608
Participants
  Number of patients undergoing ICA | 421 | 483
  Number of patients with ICA without obstructive CAD or intervention: number analyzed (Participants) | 421 | 483
  Number of patients with ICA without obstructive CAD or intervention | 119 | 223
  Number of patients with ICA without obstructive CAD: number analyzed (Participants) | 421 | 483
  Number of patients with ICA without obstructive CAD | 88 | 184
  Number of patients with ICA without intervention: number analyzed (Participants) | 421 | 483
  Number of patients with ICA without intervention | 31 | 39
Statistical Analysis 1: Comparison: CTA/CT-FFR Care Group vs Routine Clinically-indicated Diagnostic Care Group; Rate of ICA without obstructive CAD or intervention within 90 days; Test type: Other; p = 0.05, Chi-squared
Statistical Analysis 2: Comparison: CTA/CT-FFR Care Group vs Routine Clinically-indicated Diagnostic Care Group; Rate of patients underwent revascularization; Test type: Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Participant With Major Adverse Cardiovascular Event
Description: Major adverse cardiovascular event include death, myocardial infarction (MI), major complications from cardiovascular (CV) procedures or testing, and unstable angina hospitalization
Time Frame: 12 months
Population: The primary endpoint analysis was performed in both groups as the primary endpoint was assessable at baseline. However, secondary endpoints were assessed after 1-year follow-up and due to loss to follow-up（21 in CT-FFR group; 19 in standard care group）, 587 and 589 patients from each group were available for final analysis of secondary endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group
Number analyzed (Participants) | 587 | 589
Participants | 48 | 54
Statistical Analysis 1: Comparison: CTA/CT-FFR Care Group vs Routine Clinically-indicated Diagnostic Care Group; Test type: Other; p = 0.80, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.59 to 1.30]

3. Secondary Outcome: Medical Expenditure
Description: Overall cardiac medical expenditure by intention to treat at both 90 days and 12 months cumulatively
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ¥
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group
Number analyzed (Participants) | 587 | 589
¥ | 47032 (38533) | 51265 (41462)
Statistical Analysis 1: Comparison: CTA/CT-FFR Care Group vs Routine Clinically-indicated Diagnostic Care Group; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Patient Reporting Outcomes
Description: Patient reporting outcomes as measured by Seattle Angina Questionnaire-7(SAQ-7) Scale, use SAQ-7-item instrument that measures patient reported symptoms, function and quality of life for subjects with CAD within 12 months. The SAQ-7 score is calculated as the average of the physical limitation score, quality of life score and angina frequency score. The physical limitation score, quality of life score and angina frequency score range from 0 to 100 each. Therefore, the SAQ-7 score also ranges from 0 to 100.The higher the SAQ-7 socre, physical limitation score, quality of life score and angina frequency score are, the better the quality of life for patients with angina.
Time Frame: Study entry, 3 months, 6 months and12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group
Number analyzed (Participants) | 587 | 589
scores on a scale
  Seattle Angina Questionnaire-7(SAQ-7) Scale in study entry | 57.6 (4.5) | 57.4 (4.3)
  Seattle Angina Questionnaire-7(SAQ-7) Scale in 3 month | 73.8 (1.1) | 72.3 (1.0)
  Seattle Angina Questionnaire-7(SAQ-7) Scale in 6 month | 81.4 (1.3) | 80.7 (1.2)
  Seattle Angina Questionnaire-7(SAQ-7) Scale in 12 month | 86.3 (3.1) | 87 (2.9)
  Physical limitation score in study entry | 59 (4.3) | 56.9 (4.1)
  Physical limitation score in 3 month | 73 (1.1) | 70.1 (0.9)
  Physical limitation score in 6 month | 81.1 (1.7) | 79.1 (1.9)
  Physical limitation score in 12 month | 88.9 (3.3) | 88 (2.9)
  Quality of life score in study entry | 61.2 (4.7) | 62.1 (4.7)
  Quality of life score in 3 month | 77.1 (1.8) | 75 (1.9)
  Quality of life score in 6 month | 82 (1.9) | 83 (1.7)
  Quality of life score in 12 month | 87.1 (3.0) | 88.2 (3.6)
  Angina frequency score in study entry | 52.5 (4.5) | 53.2 (4.3)
  Angina frequency score in 3 month | 71.2 (1.9) | 72 (1.1)
  Angina frequency score in 6 month | 81 (1.9) | 80 (1.5)
  Angina frequency score in 12 month | 82.9 (3.0) | 84.9 (2.4)
Statistical Analysis 1: Comparison: CTA/CT-FFR Care Group vs Routine Clinically-indicated Diagnostic Care Group; Test type: Other; p = 0.15, t-test, 2 sided

5. Secondary Outcome: Cumulative Radiation Exposure
Description: Cumulative radiation exposure for any examination within 90 days and 12 months. Due to not enough data acquired, the investigators decided not to report at this time
Time Frame: 90 days, 12 months
Reporting Status: Not Posted, anticipated posting 2024-06

ADVERSE EVENTS:
Time Frame: 1 year
Description: The primary endpoint analysis was performed in both groups as the primary endpoint was assessable at baseline. However, secondary endpoints as well as adverse event were assessed after 1-year follow-up and due to loss to follow-up（21 in CT-FFR group; 19 in standard care group）, 587 and 589 patients from each group were available for final analysis of adverse event.
Arm/Group | CTA/CT-FFR Care Group | Routine Clinically-indicated Diagnostic Care Group
All-Cause Mortality (participants affected / at risk) | 2/587 | 1/589
Serious Adverse Events (participants affected / at risk) | 14/587 | 25/589
Other Adverse Events (participants affected / at risk) | 39/587 | 44/589
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTA/CT-FFR Care Group (N=587) | Routine Clinically-indicated Diagnostic Care Group (N=589)
Nonfatal myocardiol infraction (Cardiac disorders) | 7 | 9
Revascularization after 90 days (Cardiac disorders) | 7 | 16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTA/CT-FFR Care Group (N=587) | Routine Clinically-indicated Diagnostic Care Group (N=589)
Hospitalization for unstable angina (Cardiac disorders) | 39 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03901326/Prot_SAP_000.pdf